CLINICAL TRIAL: NCT03793413
Title: The Impact of Lingual Frenotomy on Bottle Feeding Mechanics: a Randomized, Controlled Trial
Brief Title: The Impact of Lingual Frenotomy on Bottle Feeding Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Responsible Party: Principal Investigator, Bobak Ghaheri, MD, Otolaryngologist, The Oregon Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ghaheri 3
Record Dates: First submitted 2018-12-29; First posted 2019-01-04 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ankyloglossia; Feeding, Bottle; Feeding Disorder of Infancy and Childhood
Keywords: tongue tie; ankyloglossia; infant feeding; bottle feeding
MeSH Terms: conditions — Ankyloglossia; Bottle Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgical group (Experimental)
  Interventions: Procedure: Lingual frenotomy
- Observation group (No Intervention)

INTERVENTIONS:
Procedure: Lingual frenotomy — A lingual frenotomy will be performed using a CO2 laser - using the NFANT bottle feeding system, the intervention arm will be compared against the observation arm to determine if there are changes in lingual mobility parameters during bottle feeding.
  Arms: Surgical group

SUMMARY:
Conservative estimates show that 3-5% of all infants have tongue tie. These studies only focus on visible, anterior tongue tie. Deeper, more visibly subtle cases of ankyloglossia have not been included in these incidence numbers, so the percentage of children with ankyloglossia is much higher than previously thought. Previous research by the investigators demonstrates that posterior tongue tie can be as problematic as anterior ties.

An available FDA-approved feeding solution allows for the measurement of infant sucking motions. This allows for detection of changes following surgical intervention. Previous ultrasound studies show the importance of the upward movement of the tongue, but further lingual movement parameters following frenotomy have not been reported.

The primary goal of this study is to record changes in lingual movement following lingual frenotomy. The investigators plan to compare improvements over time between a control, non-intervention group and a frenotomy group. Secondary goals include recording validated outcomes of reflux and feeding efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Babies who are already fully or partially bottlefeeding
* Have already worked with lactation consultant prior to appointment
* Diagnosis of tongue tie

Exclusion Criteria:

* Severe neurologic/cardiac/pulmonary comorbid diseases
* Twins/Triplets
* Other oral pathology (ie cleft lip/palate)

Ages: 3 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Improved sucking parameter on the NFANT bottle feeding system - amplitude | 10 days
  The NFANT bottle feeding system automatically generates measurements of sucking parameters. The first sucking parameter to be measured is calibrated nipple movement (amplitude)
Improved sucking parameter on the NFANT bottle feeding system - sucking frequency | 10 days
  The NFANT bottle feeding system automatically generates measurements of sucking parameters. The second sucking parameter to be measured is sucking frequency.
Improved sucking parameter on the NFANT bottle feeding system - sucking duration | 10 days
  The NFANT bottle feeding system automatically generates measurements of sucking parameters. The second sucking parameter to be measured is sucking duration.
Improved sucking parameter on the NFANT bottle feeding system - sucking smoothness | 10 days
  The NFANT bottle feeding system automatically generates measurements of sucking parameters. The second sucking parameter to be measured is sucking smoothness.

SECONDARY OUTCOMES:
Measurement of infant reflux | 10 days
  Use of a validated survey (the infant gastroesophageal reflux questionnaire revised or I-GERQ-R questionnaire). The I-GERQ-R utilizes ordinal response scales to measure the severity of symptoms associated with infant gas- troesophageal reflux disease (GERD). Scoring involves the sum- marization of 12 items (score range, 0-42), where lower scores reflect lower symptom severity.
Measurement of feeding efficiency | 10 days
  Feeding efficiency can be measured (volume of intake over measured time)

CONTACTS AND LOCATIONS:
Overall Officials: Bobak Ghaheri, MD, Principal Investigator — The Oregon Clinic
Locations (1):
- The Oregon Clinic, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Geddes DT, Langton DB, Gollow I, Jacobs LA, Hartmann PE, Simmer K. Frenulotomy for breastfeeding infants with ankyloglossia: effect on milk removal and sucking mechanism as imaged by ultrasound. Pediatrics. 2008 Jul;122(1):e188-94. doi: 10.1542/peds.2007-2553. Epub 2008 Jun 23. PMID 18573859
- [Result] Ghaheri BA, Cole M, Fausel SC, Chuop M, Mace JC. Breastfeeding improvement following tongue-tie and lip-tie release: A prospective cohort study. Laryngoscope. 2017 May;127(5):1217-1223. doi: 10.1002/lary.26306. Epub 2016 Sep 19. PMID 27641715
- [Result] Ghaheri BA, Cole M, Mace JC. Revision Lingual Frenotomy Improves Patient-Reported Breastfeeding Outcomes: A Prospective Cohort Study. J Hum Lact. 2018 Aug;34(3):566-574. doi: 10.1177/0890334418775624. Epub 2018 May 22. PMID 29787680
- [Result] Elad D, Kozlovsky P, Blum O, Laine AF, Po MJ, Botzer E, Dollberg S, Zelicovich M, Ben Sira L. Biomechanics of milk extraction during breast-feeding. Proc Natl Acad Sci U S A. 2014 Apr 8;111(14):5230-5. doi: 10.1073/pnas.1319798111. Epub 2014 Mar 24. PMID 24706845
- [Result] Capilouto GJ, Cunningham TJ, Mullineaux DR, Tamilia E, Papadelis C, Giannone PJ. Quantifying Neonatal Sucking Performance: Promise of New Methods. Semin Speech Lang. 2017 Apr;38(2):147-158. doi: 10.1055/s-0037-1599112. Epub 2017 Mar 21. PMID 28324904
- [Result] Capilouto GJ, Cunningham T, Frederick E, Dupont-Versteegden E, Desai N, Butterfield TA. Comparison of tongue muscle characteristics of preterm and full term infants during nutritive and nonnutritive sucking. Infant Behav Dev. 2014 Aug;37(3):435-45. doi: 10.1016/j.infbeh.2014.05.010. Epub 2014 Jun 20. PMID 24956503
- [Result] Capilouto GJ, Cunningham TJ. Objective assessment of a preterm infant's nutritive sucking from initiation of feeding through hospitalization and discharge. Neonatal Intensive Care. 2016 Winter;29(1):40-45. PMID 28008218